CLINICAL TRIAL: NCT06360302
Title: Contribution of Plasma Assays of Biomarkers of Muscle Metabolism During Exercise to the Assessment of Insulin Resistance in Chronic Renal Failure Patients Undergoing Hemodialysis.
Brief Title: Plasma Biomarkers of Muscle Metabolism During Exercise to the Assessment of Insulin Resistance in CKD Dialysis Patients
Acronym: KREBSome-IRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL22_0505
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Syndrome; Dialysis; Complications
Keywords: exercise test; Citric Acid Cycle; metabolomic
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise Test; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Cross-sectional comparative study with repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy volunters (Active Comparator): Voluntary participants with no chronic diseases aged 40 to 75 wishing to take part in the study and benefit from an exercise test.
  Interventions: Diagnostic Test: Exercise test; Diagnostic Test: Blood sample; Diagnostic Test: Impedancemetry
- Metabolic syndrome patients (Active Comparator): Patients aged 40 to 75 with metabolic syndrome undergoing functional assessment in the physiology department.
  Interventions: Diagnostic Test: Exercise test; Diagnostic Test: Blood sample; Diagnostic Test: Impedancemetry
- CKD dialysis patients (Experimental): Chronic renal failure patients on dialysis, stable hemodialysis for more than 3 months
  Interventions: Diagnostic Test: Exercise test; Diagnostic Test: Blood sample; Diagnostic Test: Impedancemetry

INTERVENTIONS:
Diagnostic Test: Exercise test — "Metabolic" effort test on cycloergometer with gas measurement. Gas exchanges (V'O2 and V'CO2) will be measured cycle-by-cycle using a gas analyzer connected to a flow meter Measurements will be taken every 6 minutes, at rest and during exercise on a cycloergometer, in five 6-minute increments, corresponding to intensities of 0% (rest), 20%, 30%, 40%, 50 and 60% of the subject's estimated maximum power, for a total duration of around 45 minutes.
Diagnostic Test: Blood sample — A catheter will be placed in a forearm vein to take blood samples at rest and at the end of the 5-stage stress test.
  Sampling times synchronized with stress test measurements
Diagnostic Test: Impedancemetry — measurement of anthropometric data (weight, height, waist circumference). impedancemetry will enable body composition to be analyzed by placing surface electrodes on the body. The participant will lie on an examination table and must remain at rest for 5 minutes.

SUMMARY:
This prospective, multicenter, cross-sectional, repeated-measures comparative study compared functional and biochemical response profiles to exercise between 2 groups of chronically ill patients (chronic renal failure dialysis patients and patients with metabolic syndrome) and a group of healthy subjects.

The hypothesis is that the addition of plasma metabolic intermediates associated with energy disorders linked to insulin resistance, will improve the sensitivity of the assessment of muscle oxidative metabolism abnormalities, as reported in exercise intolerant subjects.

In this way, the metabolomics approach during exercise would provide a biological and functional "signature" of insulin resistance of muscular origin, discriminating between insulin-resistant patients, healthy control subjects and dialysis patients, with an exercise metabolic profile approaching that observed in insulin-resistant patients. A better understanding of metabolic abnormalities could guide muscle rehabilitation.

Participants will be asked to perform an exercise test, with several blood samples taken at different exercise intensities.

Researchers will compare the metabolic profile of three groups: patients with chronic kidney disease, patients with metabolic syndrome and healthy subjects:

* V'O2-adjusted lactate at rest and during exercise
* The combination of exercise energy metabolism intermediates reflecting insulin resistance among Krebs cycle cofactors/substrates, ß-oxidation cofactors/substrates, amino acids

DETAILED DESCRIPTION:
Chronic renal failure (or CKD) is a chronic disease requiring end-stage replacement of renal function by extra-renal purification via hemodialysis (HD). CKD patients on dialysis suffer from numerous severe co-morbidities, limiting the possibility of renal transplantation.

Metabolic impairments are numerous and complex: dyslipidemia, phospho-calcium disorders, hormonal and nutritional disturbances.

In these patients, the onset of insulin resistance is virtually systematic, but its assessment remains a challenge. In fact, the classic screening method known as HOMA-IR, using simultaneous measurement of insulin and plasma glucose levels, is greatly affected by dialysis and the timing of its implementation. The reference method known as the hyperinsulinemic-euglycemic clamp is difficult to perform in HD patients.

While insulin resistance is a condition that can be reversed by physical activity in chronic pathologies, the absence of a validated assessment method for CKD in HD represents a missed opportunity for prevention in CKD, at a time when muscle rehabilitation programs are developing in CKD.

Moreover, insulin resistance is associated with skeletal striated muscle dysfunction in CKD patients, and constitutes another major comorbidity in these patients, as skeletal striated muscle is the main tissue utilizing glucose in response to insulin. The research team has shown that muscular dysfunctions associating reduced muscle strength and/or muscular atrophy are a morbi-mortality factor in dialysis patients. Finally, molecular abnormalities associate a switch of muscle fibers towards glycolytic fibers and mitochondrial abnormalities strongly suggesting an energy dysfunction.

In a preliminary study, the research team were able to demonstrate in dialysis patients an alteration in energy metabolism, comparable to a loss of "metabolic flexibility", mimicking that observed in insulin-resistant patients without renal dysfunction. A better understanding of the components of energy anomalies and insulin resistance could guide muscle rehabilitation protocols and prevent complications associated with insulin resistance.

Currently, the only valid, non-invasive method used in clinical practice to demonstrate impairment of muscular oxidative metabolism is the measurement of carbohydrate/lipid utilization rate during an exercise test. This "metabolic stress test" makes it possible to determine the point of maximum lipid utilization (LIPOXMAX), the current reference marker of muscle metabolism during exercise.

Nevertheless, LIPOXMAX alone cannot provide an understanding of underlying metabolic abnormalities in energy pathways, and the assay of different muscle metabolites released into plasma during exercise (and their combination) has recently emerged as a specific and early assessment of insulin resistance.

In particular, parameters such as lactate or pyruvate measured in plasma at rest have been positively correlated with the HOMA-IR index and associated with an increased risk of developing type 2 diabetes. During exercise (metabolic stress test), lactate levels in insulin-resistant patients differ from those in healthy controls.

In view of the abnormalities of oxidative muscle metabolism in CKD and insulin-resistant patients, the measurement of lactate at rest and during exercise, adjusted for V'O2, could reveal a profile enabling discrimination of CKD and insulin-resistant patients from healthy control subjects.

With the addition of plasma metabolic intermediates associated with energy disorders linked to insulin resistance, The investigators hypothesize that their measurement during exercise will improve the sensitivity of the assessment of muscle oxidative metabolism abnormalities, as reported in exercise-intolerant subjects.

The metabolomics approach during exercise would provide a biological and functional "signature" of muscle-induced insulin resistance in haemodialysis patients. A better understanding of metabolic abnormalities could guide muscle rehabilitation.

This prospective, cross-sectional, repeated-measures comparative study comparing functional and biochemical response profiles to exercise between 2 groups of chronically ill patients and a group of healthy subjects.

This comparison of the metabolisms of the 3 groups is analyzed using repeated plasma sampling at different effort intensities.

* Plasma lactate adjusted to V'O2 (ratio) at rest and during exercise.
* V'O2-adjusted metabolic profile at rest and during exercise through a combination of exercise energy metabolism intermediates based on candidate metabolites with a significant correlation coefficient >0.7 compared to LIPOXmax and/or HOMA-IR, among the following:
* Krebs cycle cofactors/substrates (lactate, pyruvate, malate, citrate, succinate, fumarate and alpha-cetoglutarate)
* ß-oxidation cofactors/substrates (free fatty acids, acyl-carnitine profile, beta-hydroxybutyrate, acetoacetate)
* Amino acid profile
* Acyl carnitine profile

ELIGIBILITY:
Inclusion Criteria:

Group 1: Healthy subjects:

* Postmenopausal women aged 40 to 75 or men aged 40 to 75
* No chronic disease or treatment
* BMI <30 kg/m², or
* Fasting blood glucose < 1.10 g/dL

Group 2: metabolic syndrome patients

* Postmenopausal women aged 40 to 75 or men aged 40 to 75
* Metabolic syndrome as defined by the International Diabetes Federation (IDF 2006)5
* BMI <30 kg/m² and waist circumference >80 cm for women and >94 cm for men
* Insulin resistance defined by HOMA-IR>2.4

Group 3: CKD dialysis patients

* Non-diabetics
* Postmenopausal women aged 40 to 75 and men aged 40 to 75
* BMI <30 kg/m².
* Chronic kidney disease patients on dialysis - stable on HD for more than 3 months

Patients and healthy subjects will be matched on age (+/-3 years) and sex

Exclusion Criteria:

* Non-stabilized pathology incompatible with physical exercise
* Ongoing exercise retraining program
* Nutritional supplementation in the 4 weeks preceding the study (antioxidants, vitamins, etc.)
* Treatment influencing mitochondrial function (metformin, statin, etc.)
* Failure to obtain written informed consent after a period of reflection
* Subject not affiliated to a social security scheme, or not benefiting from such a scheme.
* Person protected by law (under guardianship or curatorship)
* Patient deprived of liberty
* Diabetic patient
* Family dyslipidemia
* Participants who have reached the maximum amount of compensation for their participation in research projects
* Person under psychiatric care
* Person participating in another research project with an exclusion period still in progress.
* Mentally handicapped, dementia, illiterate, language barrier with inability to understand study purpose and methodology

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
Compare V'O2-adjusted plasma lactate profile at rest and during exercise (metabolic stress test), between chronic renal failure patients, patients with metabolic syndrome and healthy subjects. | Baseline (rest), 6, 12, 18, 24, 30 minutes
  Measurements will be taken every 6 minutes, at rest and during exercise on a cycloergometer, corresponding to intensities of 0% (rest) 20%, 30%, 40%, 50 and 60% of the subject's estimated maximum power.
  The gas exchange measurement (V'O2 and V'CO2 (milliliter per minute mL/min)) will be carried out cycle-by-cycle using a gas analyzer connected to a flow meter.
  The intensity corresponding to the rate of maximum lipid oxidation will be defined as LIPOXMAX, and will be expressed in Watts (W), and as a % of theoretical VO2max.
  Carbohydrate (G) and lipid (L) oxidation rates will be calculated as follows:
  * G (mg/min) = 4.585 VCO2 - 3.2255 VO2
  * L (mg/min) = 1.6946 VO2 - 1.7012 VCO2
  Blood sampling at various levels on a peripheral venous catheter synchronized with stress test measurements.
  A comparison will be made on the basis of an analysis of variance by ANOVA one way after verification of the conditions of application or a rank test by analysis via Kruskal-Wallis.

SECONDARY OUTCOMES:
Compare between the 3 groups their metabolic profile (Krebs cycle cofactors/substrates) adjusted to V'O2 at rest and during exercise. | Baseline (rest), 6, 12, 18, 24, 30 minutes
  "Metabolic" Exercice test on a cycloergometer with gas measurement and peripheral venous sampling at various intensities.
  HOMA-IR score (Homeostatic model assessment of insulin resistance) is calculated using simultaneous measurement of insulin and plasma glucose levels, a score above 2.4 is diagnostic of insulin resistance.
  A combination of exercise energy metabolism intermediates based on candidate metabolites with a significant correlation coefficient >0.7 compared to LIPOXmax and/or HOMA-IR, from among the following Krebs cycle cofactors/substrates : lactate, pyruvate, malate, citrate, succinate, fumarate and alpha-cetoglutarate
  Correlations will be characterized by Pearson's correlation test (correlation considered significant for coefficients >0.7).
  Logistic regression analysis will be used to characterize insulin resistance in the different groups on the basis of the data collected.
Compare between the 3 groups their metabolic profile (ß-oxidation cofactors/substrates) adjusted to V'O2 at rest and during exercise. | Baseline (rest), 6, 12, 18, 24, 30 minutes
  "Metabolic" Exercise test on a cycloergometer with gas measurement and peripheral venous sampling at various intensities.
  HOMA-IR score (Homeostatic model assessment of insulin resistance) is calculated using simultaneous measurement of insulin and plasma glucose levels, a score above 2.4 is diagnostic of insulin resistance.
  A combination of exercise energy metabolism intermediates based on candidate metabolites with a significant correlation coefficient >0.7 compared to LIPOXmax and/or HOMA-IR, from among the following ß-oxidation cofactors/substrates : free fatty acids, acyl-carnitine profile, beta-hydroxybutyrate, acetoacetate
  Correlations will be characterized by Pearson's correlation test (correlation considered significant for coefficients >0.7).
  Logistic regression analysis will be used to characterize insulin resistance in the different groups on the basis of the data collected.
Compare between the 3 groups their metabolic profile (amino acids) adjusted to V'O2 at rest and during exercise. | Baseline (rest), 6, 12, 18, 24, 30 minutes
  "Metabolic" Exercise test on a cycloergometer with gas measurement and peripheral venous sampling at various intensities.
  HOMA-IR score (Homeostatic model assessment of insulin resistance) is calculated using simultaneous measurement of insulin and plasma glucose levels, a score above 2.4 is diagnostic of insulin resistance.
  A combination of exercise energy metabolism intermediates based on candidate metabolites with a significant correlation coefficient >0.7 compared to LIPOXmax and/or HOMA-IR, from among the following amino acids.
  Correlations will be characterized by Pearson's correlation test (correlation considered significant for coefficients >0.7).
  Logistic regression analysis will be used to characterize insulin resistance in the different groups on the basis of the data collected.
Compare between the 3 groups their metabolic profile (acyl-carnitine profiles) adjusted to V'O2 at rest and during exercise. | Baseline (rest), 6, 12, 18, 24, 30 minutes
  "Metabolic" Exercise test on a cycloergometer with gas measurement and peripheral venous sampling at various intensities.
  HOMA-IR score (Homeostatic model assessment of insulin resistance) is calculated using simultaneous measurement of insulin and plasma glucose levels, a score above 2.4 is diagnostic of insulin resistance.
  A combination of exercise energy metabolism intermediates based on candidate metabolites with a significant correlation coefficient >0.7 compared to LIPOXmax and/or HOMA-IR, from among the following acyl-carnitine profiles
  Correlations will be characterized by Pearson's correlation test (correlation considered significant for coefficients >0.7).
  Logistic regression analysis will be used to characterize insulin resistance in the different groups on the basis of the data collected.
Anthropometry Comparison between the 3 groups | Baseline (rest)
  calculation of BMI with the Measurement of weight (in kilograms Kg) and height (in centimetres cm).

CONTACTS AND LOCATIONS:
Overall Officials: GRILLET Pierre-Edouard, Pharma D. PhD, Study Director — University Hospital, Montpellier
Locations (2):
- France (2):
  - AIDER Santé Fondation Charles Mion Montpellier, site Lapeyronie, Montpellier
  - Montpellier University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No